CLINICAL TRIAL: NCT03758807
Title: A Follow-up Comparison of Active Versus Passive Manual Therapy in Patients With Low Back Pain: a Randomized Control Trial
Brief Title: A Follow-up Comparison of Active Versus Passive Manual Therapy in Patients With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Ambrose University (Other)
Responsible Party: Principal Investigator, Kevin Farrell, Professor, Chair of Clinical Residency Program in Orthopaedic Physical Therapy, St. Ambrose University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: StAmbroseUactive passive
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2018-11

CONDITIONS: Low Back Pain; Manual Therapy; Education
Keywords: Low back pain; Manual Therapy; Education; Neuroplasticiy
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant
Masking Description: Patients were randomly assigned to one of two treatment groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive treatment (Sham Comparator): Passive treatment will consist of Manual Therapy with biomechanical explanation of the technique.
  Interventions: Other: Manual Therapy with Traditional Biomechanical Explanation
- Active Treatment (Experimental): Active treatment will consist of Manual Therapy with a neuroplasticity explanation of the technique.
  Interventions: Other: Manual Therapy with Neuroplastiicity Explanation

INTERVENTIONS:
Other: Manual Therapy with Traditional Biomechanical Explanation — Patients will lie prone and receive lumbar Posterior to Anterior (AP) Pressure with a traditional biomechanical or anatomic explanation of the technique..
  Arms: Passive treatment
Other: Manual Therapy with Neuroplastiicity Explanation — Patients will lie prone and receive lumbar Posterior to Anterior (PA) Pressure with a neuroplastic explanation of the technique.
  Arms: Active Treatment

SUMMARY:
To determine if there is any carry over difference between the type of education provided about common treatment techniques for patients with low back pain. This will be looked at right after treatment and when patients return on their second visit after they do a common exercise program for a few days.

DETAILED DESCRIPTION:
Prior clinical trials have shown that patients respond differently to different explanations about interventions performed. A recent randomized clinical trial demonstrated that a 10-minute manual therapy treatment (prone lumbar Posterior to Anterior mobilization (PA's) with a neuroplasticity vs. traditional biomechanical explanation) produced an immediate, significant improvement in straight leg raise (SLR) and pain for patients with chronic low back pain. However, there is a need to examine whether there is any carry over (48-96 hours) or if utilizing a home exercise program (HEP), aimed at increasing the various sensory process applied in the clinic, produces any carry over. This will be looked at in patients with who are provided different explanations about common back treatment techniques to see if there will be any change in pain rating or back and leg movement.

ELIGIBILITY:
Inclusion Criteria:

* adults over the age of 18
* patients presenting at PT with a primary complaint of LBP
* LBP being present for 6 months or more
* fluent in English
* willing to participate in the study.

Exclusion Criteria:

* under age 18
* not able to read/understand the English language
* prisoners
* no medical issues precluding physical therapy treatment (red flags)
* no medical precautions to the use of manual therapy (metal, skin lesions, etc.)
* prior spine surgery
* unable to lay prone for the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Low Back Pain Rating | Change from baseline to initial treatment
  Numeric Pain Rating Scale for Back Pain (0 = no pain and 10 = worst pain). The minimal detectable change (MDC) for the NPRS for low back pain is reported to be 2.0.
  LBP is reported to be 2.0.
Low Back Pain Rating | Change from initial treatment to 2-4 days
  Numeric Pain Rating Scale for Back Pain (0 = no pain and 10 = worst pain). The minimal detectable change (MDC) for the NPRS for low back pain is reported to be 2.0.
Lumbar flexion | Change from baseline to initial treatment
  Active trunk forward flexion in cm (distance finger tips to floor)
Lumbar flexion | Change from initial treatment to 2-4 days
  Active trunk forward flexion in cm (distance finger tips to floor)
Straight Leg Raise | Change from baseline to initial treatment
  Neurodynamic Measurement of Leg Raise (lower limb tension test)
Straight Leg Raise | Change from initial treatment to 2-4 days
  Neurodynamic Measurement of Leg Raise (lower limb tension test)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Farrell, Principal Investigator — St. Ambrose University
Locations (1):
- Kevin Farrell, Davenport, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Louw A, Farrell K, Wettach L, Uhl J, Majkowski K, Wedling M. Immediate effects of sensory discrimination for chronic low back pain: a case series. New Zealand Journal of Physiotherapy. 2015;43(2):58-63.
- [Result] Louw A, Farrell K, Landers M, Barclay M, Goodman E, Gillund J, McCaffrey S, Timmerman L. The effect of manual therapy and neuroplasticity education on chronic low back pain: a randomized clinical trial. J Man Manip Ther. 2017 Dec;25(5):227-234. doi: 10.1080/10669817.2016.1231860. Epub 2016 Sep 22. PMID 29449764